CLINICAL TRIAL: NCT05591612
Title: Increasing Vegetable Intake Using Monosodium Glutamate: A Reduced-Effort Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: American Society for Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-396
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Healthy Nutrition; Culinary Medicine; Sodium Excess
MeSH Terms: conditions — Hypernatremia | interventions — Salts; Sodium Glutamate; Sodium Chloride; Sodium Chloride, Dietary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 50% NaCl and 50% MSG Seasoning Mix (Experimental): Participants received cooking demonstrations and nutrition education, and were asked to use the seasoning provided (50% NaCl and 50% MSG Seasoning Mix) on vegetables and foods prepared. Then they recorded their food intake to compare vegetable intake to other groups.
  Interventions: Behavioral: Salt replacement seasoning (50% salt and 50% MSG) mix
- 70% NaCl and 30% MSG Seasoning Mix (Experimental): Participants received cooking demonstrations and nutrition education, and were asked to use the seasoning provided (70% NaCl and 30% MSG Seasoning Mix) on vegetables and foods prepared. Then they recorded their food intake to compare vegetable intake to other groups.
  Interventions: Behavioral: Salt replacement seasoning (70% salt and 30% MSG) mix
- NaCl seasoning (Experimental): Active Control Participants received cooking demonstrations and nutrition education, and were asked to use table salt on vegetables and foods prepared. Then they recorded their food intake to compare vegetable intake to other groups.
  Interventions: Behavioral: NaCl (sodium chloride/table salt)

INTERVENTIONS:
Behavioral: Salt replacement seasoning (50% salt and 50% MSG) mix — Individuals in this group were provided a seasoning that replaced 50 % regular salt with a reduced-sodium MSG substitute. This study assessed the vegetable intake using the intervention of 50/50 MSG Mix to be added to vegetables in diet.
  Arms: 50% NaCl and 50% MSG Seasoning Mix
Behavioral: Salt replacement seasoning (70% salt and 30% MSG) mix — Individuals in this group were provided a seasoning that replaced 30 % regular salt with a reduced-sodium MSG substitute. This study assessed the vegetable intake using the intervention of 70/30 MSG Mix to be added to vegetables in diet.
  Arms: 70% NaCl and 30% MSG Seasoning Mix
Behavioral: NaCl (sodium chloride/table salt) — Individuals in this group were asked to use normal seasoning of regular salt. This study assessed the vegetable intake using table salt to be added to vegetables in diet.
  Arms: NaCl seasoning

SUMMARY:
Food Intake Study: This will be a 4-week randomized controlled intervention study with a vegetable intake questionnaire, daily food intake, and seasoning usage measurement to test the acceptability of different seasoning ingredients and vegetable intake in healthy adults. Participants will be randomly assigned to one of three groups (a) vegetables prepared with 50% NaCl and 50% MSG (50/50MSG Mix); (b) vegetables prepared with 70% NaCl and 30% MSG (70/30 MSG Mix); (c) vegetables prepared with NaCl (table salt).

Sensory Evaluation Study: A sensory evaluation utilizing all seasoning methods from the intervention will be conducted at a Texas Tech University culinary education lab. In a Texas Tech University culinary education lab, 2-4 vegetables will be cooked and seasoned with either 50/50MSG Mix, 70/30 MSG Mix, or NaCl for taste testing. Then, using a standardized form, participants will rate their acceptability and preference of each vegetable, including sensory characteristics such as appearance, color, odor, texture, and flavor.

DETAILED DESCRIPTION:
Food Intake Study: This will be a 4-week randomized controlled intervention study with a vegetable intake questionnaire, daily food intake, and seasoning usage measurement to test the acceptability of different seasoning ingredients and vegetable intake in healthy adults. Participants will be randomly assigned to one of three groups (a) vegetables prepared with 50% NaCl and 50% MSG (50/50MSG Mix); (b) vegetables prepared with 70% NaCl and 30% MSG (70/30 MSG Mix); (c) vegetables prepared with NaCl (table salt). Before the intervention, each group will be asked to keep a daily food intake record for one week to determine baseline vegetable intake. Each group will receive a culinary medicine program electronically, including recipe demonstrations, cooking skills, and nutrition education videos to provide instruction for vegetable consumption according to the Dietary Guidelines for Americans. According to each treatment group, a bottle of seasoning ingredients will be provided to use on vegetables. Prior to the intervention, participants will be 1) instructed on how to track daily food intake data using the MyFitnessPal® app, 2) track food intake for seven days, and 3) complete a questionnaire regarding vegetable intake pre-intervention. According to the group assignment, each treatment group will also receive a bottle of a seasoning blend that includes either 50/50MSG Mix, 70/30 MSG Mix, or NaCl to use on vegetables prepared at home. According to the Dietary Guidelines for Americans, culinary medicine education (recipe demonstrations, cooking skills, and education videos for vegetable consumption) will be delivered electronically at baseline and once per week for four weeks to each participant. For four weeks, participants will track all meals daily, including vegetables prepared with designated seasoning at home. Remote follow-ups and dietary intake will be conducted weekly. After the intervention, the participants will 1) complete the same vegetable intake questionnaire for the four weeks of the intervention and 2) return the bottle of seasoning blend provided. Usage of seasoning for four weeks will be recorded. Data analyses will evaluate the changes in outcomes within and between groups. Participants will also be informed of the sensory evaluation study to be included among other participants of that study. MSG_Diet Food Questionaries (Updated).docx MyFitness Pal instructions.docx

Sensory Evaluation Study: A sensory evaluation utilizing all seasoning methods from the intervention will be conducted at a Texas Tech University culinary education lab. In a Texas Tech University culinary education lab, 2-4 vegetables will be cooked and seasoned with either 50/50MSG Mix, 70/30 MSG Mix, or NaCl for taste testing. Then, using a standardized form, participants will rate their acceptability and preference of each vegetable, including sensory characteristics such as appearance, color, odor, texture, and flavor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above

Exclusion Criteria:

* Allergy or aversion to MSG (monosodium glutamate) or potassium chloride
* Those that do not have a smart phone with the ability to download an app.
* Those who do not have a full kitchen and the willingness and ability to prepare vegetables according to a recipes.
* Those with an allergy, aversion, or dislike to vegetables that would make them not consume any vegetables during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Vegetable Intake | 5 weeks
  To assess the consumption of vegetables by the participant measured by data from self-recorded diet as entered in smart phone application (My Fitness Pal©).

SECONDARY OUTCOMES:
Vegetable Palatability | day one (15 minutes)
  Preference Test
  Preference Test Scale
  * Scale Title: Likert Scale for Vegetable Preference
  * Minimum Value: 1 (indicating "dislike extremely")
  * Maximum Value: 9 (indicating "like extremely")
  * Higher Scores Indicate: A better outcome, meaning higher scores reflect a greater preference for the vegetables seasoned with the various NaCl/MSG mixtures.
Vegetable Palatability | day one (15 minutes)
  Triangle Sensory Evaluation Test
  Triangle Test Scale
  * Scale Title: Confidence Scale for Triangle Test
  * Minimum Value: 1 (indicating "not confident")
  * Maximum Value: 5 (indicating "completely confident")
  * Higher Scores Indicate: A better outcome in terms of confidence level in identifying the odd sample out. Higher scores reflect greater confidence in distinguishing between the NaCl/MSG mixtures and pure NaCl.
Seasoning Usage | 5 weeks
  Determine which group used the most seasoning Each group will be provided a bottle of seasoning. It will be weighed prior to them taking the seasoning. The participants will be asked to bring the remaining seasoning back to weight to determine the amount of seasoning usage during the 4 week study.
  Usage of seasoning for four weeks will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Galyean, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Nutrition and Metabolic Health Initiative, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maher C, Alcorn M, Childress A, Dawson JA, Galyean S. Increasing Vegetable Intake Using Monosodium Glutamate in a Randomized Controlled Trial: A Culinary Medicine Intervention. Food Sci Nutr. 2025 Jun 17;13(6):e70441. doi: 10.1002/fsn3.70441. eCollection 2025 Jun. PMID 40535918